CLINICAL TRIAL: NCT06876220
Title: The Role of Anchoring and Distraction in the Effectiveness of Mindfulness on Reducing Emotional Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Shui-fong, Director, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHongKong(JC PandA_fMRI)
Record Dates: First submitted 2023-11-26; First posted 2025-03-14 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Issue; Emotional Adjustment
Keywords: mindfulness; emotion regulation; emotion care; distraction; anchoring
MeSH Terms: conditions — Emotional Regulation | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Two-armed, waitlist randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Participants will receive an 8-week mindfulness-based group intervention, namely Mindfulness-based Cognitive Therapy for Life (MBCT-L).
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy for Life (MBCT-L)
- waitlist controlled group (No Intervention): Participants in the wait-list control group will receive the same intervention, two months after the experimental group completed the intervention.

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy for Life (MBCT-L) — MBCT-L is an 8-week group intervention where participants are guided to practice mindfulness and cognitive exercise. The course covers themes such as anchoring, acceptance, and decentering. The course will be provided by mindfulness teachers who have completed the training offered by Oxford Mindfulness Foundation (OMF). Throughout the eight weeks, the course guides the participants through various themes such as anchoring, acceptance, and decentering. The sessions involve guided mindfulness practices, reflection, discussion, inquiry, and weekly home practice. The language of instruction is Cantonese.
  Arms: intervention group

SUMMARY:
The current study aims to investigate the effectiveness of the 8-week Mindfulness-Based Cognitive Therapy for Life (MBCT-L) on the use of anchoring and distraction as emotion care/regulation strategies. It is hypothesized that anchoring and distraction are related but different processes, which could be evidenced by fMRI. The investigators further hypothesized that mindfulness training could lead to functional changes in the brain, which could also be evidenced by fMRI.

DETAILED DESCRIPTION:
To test the hypotheses, the participants will be randomly allocated to either the experimental group or the waitlist control group. Both groups will complete behavioral measures and an fMRI experiment before the experimental group's intervention (T0). The experimental group will receive Mindfulness-Based Cognitive Therapy for Life (MBCT-L) between T0 and T1, while the waitlist control will receive no treatment during this period. Both groups will complete the behavioral measures and the fMRI experiment again after the experimental group finishes the MBCT-L course (T1).

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Currently registered in post-graduated program with professional counselling training

Exclusion Criteria:

* History of neurological or other disorders affecting the brain (such as encephalitis, epilepsy, birth defects, or polio)
* Have experienced a concussion, head or brain trauma, seizures, loss of consciousness
* Have been injured in the eye by a metallic foreign body.
* Have been injured by metallic foreign body (e.g. bullet, shrapnel)
* History of sickle cell anemia/kidney disease/diabetes, asthma, or allergies
* Long-term use of medication is required
* Currently pregnant or breast feeding.
* Had the following conditions or implants in their body:

  * Surgical clips
  * Cardiac pacemaker
  * Neurostimulator/internal electrodes
  * Insulin pump
  * Internal shunt
  * Metal screen / suture
  * Cochlear implants
  * Hearing aid
  * Eye implants/eyelid springs
  * Orthopaedic devices (e.g. pins, nails, screws)
  * Prosthetic heart valve
  * Breast tissue expander
  * Tattoo or permanent eye-lining
  * Body ring
  * Patch/Blood Glucose Monitor
  * Dentures
  * Intrauterine contraceptive device
  * Metal blockage in the blood vessel/metal foreign body in the body

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Brain activation during the emotion care/regulation task | Baseline (2 weeks before the intervention), Post-intervention (14-16 weeks after baseline)
  BOLD signal contrast when the participants performing an emotion counting Stroop task.
Reaction time during the emotion care/regulation task | Baseline (2 weeks before the intervention), Post-intervention (14-16 weeks after baseline)
  Reaction time of the correct response in the emotion counting Stroop task.
Accuracy during the emotion care/regulation task | Baseline (2 weeks before the intervention), Post-intervention (14-16 weeks after baseline)
  Accuracy of the emotion counting Stroop task.
Mindfulness | Baseline (2 weeks before the intervention), Post-intervention (14-16 weeks after baseline), Follow-up (22-24 weeks after baseline)
  The mean score of Cognitive and Affective Mindfulness Scale-Revised (CAMS-R, Feldman, Hayes, Kumar, Greeson, & Laurenceau, 2007) is a self-report 5-point Likert scale measuring individual differences in mindfulness that includes 12 items. The mean score ranged from 1 to 5. A higher score means a higher level of mindfulness, i.e. an expected outcome from an effective mindfulness intervention.
Psychological well-being | Baseline (2 weeks before the intervention), Post-intervention (14-16 weeks after baseline), Follow-up (22-24 weeks after baseline)
  The mean score of Psychological Well-being Scale (PWBS; Ryff et al., 1995) includes 18 items measuring 6 aspects of wellbeing and happiness: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Participants used a 5-point Likert scale, ranging from 1 = highly disagree to 5 = highly agree, to rate the 18 statements. The mean score ranged from 1 to 5. A higher score means a higher level of psychological well-being, i.e. an expected outcome from an effective mindfulness intervention.
Use of distraction as a emotion care/regulation strategy | Baseline (2 weeks before the intervention), Post-intervention (14-16 weeks after baseline), Follow-up (22-24 weeks after baseline)
  The mean scores of five items of the self-developed scale to assess the use of distraction and its connection to attentional deployment with a pilot test. Participants used a 5-point Likert scale, ranging from 1 = never to 5 = always, to rate the five statements. The mean score ranged from 1 to 5. A higher score indicates a greater tendency to employ distraction as an emotion regulation strategy. It's important to note that the score only reflects the habitual usage of this strategy and does not imply a better or worse outcome.
Use of anchoring as a emotion care/regulation strategy | Baseline (2 weeks before the intervention), Post-intervention (14-16 weeks after baseline), Follow-up (22-24 weeks after baseline)
  The mean score of five items of the self-developed scale to assess the use of anchoring with a pilot test. Participants used a 5-point Likert scale, ranging from 1 = never to 5 = always, to rate the five statements. The mean score ranged from 1 to 5. A higher score indicates a greater tendency to employ distraction as an emotion regulation strategy. It's important to note that the score only reflects the habitual usage of this strategy and does not imply a better or worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shui-fong Lam, PhD, Study Director — The University of Hong Kong; Gloria HY Wong, Principal Investigator — The University of Hong Kong
Locations (1):
- Jockey Club "Peace and Awareness" Mindfulness Culture in Schools Initiative, Faculty of Social Sciences, The University of Hong Kong, Hong Kong, Hong Kong